CLINICAL TRIAL: NCT06104839
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase 2a Study to Evaluate the Efficacy and Safety of NXC736 in Patients with Moderate and Severe Alopecia Areata
Brief Title: Safety and Efficacy of Oral NXC-736 in Adult Participants with Moderate and Severe Alopecia Areata
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NEXTGEN Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NXC736-101
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NXC736 (Experimental)
  Interventions: Drug: NXC736
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NXC736 — oral administration
  Arms: NXC736
Drug: Placebo — oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of NXC-736 monotherapy in participants with severe alopecia areata (AA).

ELIGIBILITY:
Inclusion Criteria:

* Men or women between ≥19 and ≤65 years of age at the time of informed consent
* Moderate and severe alopecia areata as assessed by a SALT score of 25% ≤ SALT < 95% at Screening and Day 1/Baseline
* Current episode of hair loss for ≥6 months but <8 years
* Stable disease condition (no significant growth of hair) in the last 6 months as assessed by the Investigator
* Willing to keep the same hair style and color (eg, hair products, process, and timing for hair appointments) for the duration of the study

Exclusion Criteria:

* Participants with the following medical history confirmed during screening:

  * ohter Types of alopecia other than alopecia areata (such as cicatricial/scarring alopecia [including central centrifugal cicatricial alopecia], traction alopecia, androgenic alopecia, telogen effluvium, etc.)
* Active scalp inflammation, scalp infection, scalp psoriasis, or any other scalp condition that may interfere with the SALT assessment
* Previous use of Janus kinase (JAK) inhibitor (oral or topical), including participation in clinical studies of JAK inhibitors

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — check the ID card
Enrollment: 96 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-24 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change(%) in SALT score from baseline at Week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital., Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul

IPD SHARING:
Plan to Share IPD: No